CLINICAL TRIAL: NCT00160524
Title: A Phase III Multi-national, Multi-centre, Open Label, Safety Study to Assess the Safety of Chronic Therapy With the Humanised Anti-TNF PEG Conjugate CDP870 400 mg sc, (Dosed 4-weekly), in the Treatment of Patients With Active Crohn's Disease Who Have Previously Completed Studies CDP870-031 or CDP870-032
Brief Title: A follow-on Safety Study of CDP870 in Subjects With Crohn's Disease (CD) Who Have Completed a 26-week Double Blind Study CDP870-031 [NCT00152490] or CDP870-032 [NCT00152425]
Acronym: PRECiSE 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C87033; 2005-002622-60 (EudraCT Number)
Expanded Access: NCT03559660 (No longer available)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2013-10-10 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2013-08

CONDITIONS: Crohn's Disease
Keywords: Certolizumab Pegol; Cimzia; CDP870; CZP
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Certolizumab Pegol (Experimental): 400 mg subcutaneous injection every 4 weeks from Week 2 to Week 362.
  Interventions: Biological: Certolizumab Pegol (CDP870)

INTERVENTIONS:
Biological: Certolizumab Pegol (CDP870) — Liquid for subcutaneous injection, 200 mg/ml. 400 mg at Week 2, and every 4 weeks thereafter until Week 362. Up to 84 months of therapy in this study.
  Other Names: Cimzia; CDP870; CZP

SUMMARY:
An open-label follow-on safety study of CDP870 (400 mg every 4 weeks) in patients with Crohn's Disease who have completed a 26-week blinded study (CDP870-031 [NCT00152490] or CDP870-032 [NCT00152425]).

ELIGIBILITY:
Inclusion Criteria:

* Participation in either of the CDP870-031 [NCT00152490] or CDP870-032 [NCT00152425] clinical studies in which the subject completed the trial at Week 26. Subjects may have received active or placebo or both treatments in the prior study
* Subjects must be able to understand the information provided to them and give written informed consent

Exclusion Criteria:

* Any exclusion criterion that would have prevented the subject's participation in the qualifying pivotal study CDP870-031 [NCT00152490] or CDP870-032 [NCT00152425], although the criterion that excludes previous participation in a clinical trial of Certolizumab Pegol does not apply. In addition there are no limits on the Clinical Disease Activity Index (CDAI) score at entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2004-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (206):
- United States (47):
  - 45102, Birmingham, Alabama
  - 45028, Huntsville, Alabama
  - 45144, Tucson, Arizona
  - 45095, Orange, California
  - 45006, San Diego, California
  - 45131, San Diego, California
  - 45130, Colorado Springs, Colorado
  - 45094, Gainesville, Florida
  - 45029, Jacksonville, Florida
  - 45087, Miami, Florida
  - 45085, Plantation, Florida
  - 45143, Atlanta, Georgia
  - 45064, Savannah, Georgia
  - 45138, Columbus, Indiana
  - 45111, Louisville, Kentucky
  - 45105, Annapolis, Maryland
  - 45033, Chevy Chase, Maryland
  - 45013, Laurel, Maryland
  - 45057, Plymouth, Minnesota
  - 45108, Jefferson City, Missouri
  - 45031, Lincoln, Nebraska
  - 45035, Berlin, New Jersey
  - 45124, Florham Park, New Jersey
  - 45018, New Brunswick, New Jersey
  - 45009, Great Neck, New York
  - 45070, New York, New York
  - 45117, Rochester, New York
  - 45003, Raleigh, North Carolina
  - 45040, Winston-Salem, North Carolina
  - 45081, Cincinnati, Ohio
  - 45091, Cincinnati, Ohio
  - 45054, Dayton, Ohio
  - 45039, Oklahoma City, Oklahoma
  - 45041, Tulsa, Oklahoma
  - 45048, Portland, Oregon
  - 45084, Chattanooga, Tennessee
  - 45113, Germantown, Tennessee
  - 45071, Nashville, Tennessee
  - 45119, Nashville, Tennessee
  - 45022, Houston, Texas
  - 45073, San Antonio, Texas
  - 45020, Salt Lake City, Utah
  - 45139, Salt Lake City, Utah
  - 45052, South Ogden, Utah
  - 45078, Christiansburg, Virginia
  - 45109, Norfolk, Virginia
  - 45135, Tacoma, Washington
- Australia (14):
  - 11001, Adelaide
  - 11016, Ballarat
  - 11011, Bankstown
  - 11007, Box Hill
  - 11013, Frankston
  - 11010, Fremantle
  - 11015, Garran
  - 11017, Herston
  - 11014, Lauceston
  - 11003, Melbourne
  - 11004, Melbourne
  - 11005, New Lambton
  - 11018, Newtown
  - 11012, Parkville
- Austria (3):
  - 46005, Graz
  - 46006, Linz
  - 46002, Vienna
- Belarus (3):
  - 12001, Minsk
  - 12003, Minsk
  - 12002, Vitebsk
- Belgium (3):
  - 13004, Brussels
  - 13001, Ghent
  - 13002, Liège
- Bulgaria (2):
  - 15001, Sofia
  - 15002, Sofia
- Canada (5):
  - 16014, Halifax
  - 16021, Ottawa
  - 16013, Toronto
  - 16001, Vancouver
  - 16010, Vancouver
- Czechia (11):
  - 18003, Brno
  - 18011, České Budějovice
  - 18006, Hradek Kralove
  - 18009, Mělník
  - 18007, Olomouc
  - 18008, Olomouc
  - 18010, Pardubice
  - 18005, Plzen - Lochotin
  - 18002, Prague
  - 18004, Prague
  - 18012, Prague
- Denmark (8):
  - 19004, Aalborg
  - 19002, Aarhus
  - 19008, Copenhagen
  - 19009, Copenhagen
  - 19001, Glostrup Municipality
  - 19010, Herlev
  - 19007, Hvidovre
  - 19005, Odense C
- Estonia (2):
  - 20001, Tallinn
  - 20002, Tartu
- 48001, Tbilisi, Georgia
- Germany (13):
  - 22002, Berlin
  - 22006, Berlin
  - 22009, Berlin
  - 22021, Cologne
  - 22026, Dresden
  - 22013, Göttingen
  - 22017, Hanover
  - 22015, Kiel
  - 22024, Leipzig
  - 22003, Magdeburg
  - 22001, Minden
  - 22008, Münster
  - 22005, Wilhelmshaven
- 23002, Shatin, Hong Kong
- Hungary (11):
  - 24002, Budapest
  - 24012, Budapest
  - 24015, Budapest
  - 24001, Debrecen
  - 24014, Dunaújváros
  - 24010, Győr
  - 24005, Gyula
  - 24009, Pécs
  - 24008, Szeged
  - 24011, Szekszárd
  - 24007, Veszprém
- Israel (3):
  - 26004, Beersheba
  - 26007, Haifa
  - 26006, Jerusalem
- Italy (5):
  - 27002, Bologna
  - 27001, Milan
  - 27004, Palermo
  - 27006, Roma
  - 27007, Roma
- Latvia (2):
  - 28001, Riga
  - 28003, Riga
- 29001, Kaunas, Lithuania
- New Zealand (5):
  - 31002, Auckland
  - 31001, Christchurch
  - 31005, Hamilton
  - 31003, Tauranga
  - 31004, Tauranga
- Norway (5):
  - 32009, Hamar
  - 32001, Haugesund
  - 32005, Oslo
  - 32008, Oslo
  - 32004, Tromsø
- Poland (16):
  - 33022, Bialystok
  - 33004, Bydgoszcz
  - 33002, Krakow
  - 33010, Krakow
  - 33011, Lodz
  - 33012, Lodz
  - 33019, Lublin
  - 33020, Opole
  - 33003, Sopot
  - 33013, Szczecin
  - 33001, Warsaw
  - 33007, Warsaw
  - 33009, Warsaw
  - 33016, Warsaw
  - 33006, Wroclaw
  - 33021, Wroclaw
- Russia (9):
  - 34017, Lipetsk
  - 34006, Moscow
  - 34015, Moscow
  - 34016, Nizhny Novgorod
  - 34001, Saint Petersburg
  - 34005, Saint Petersburg
  - 34007, Saint Petersburg
  - 34013, Saint Petersburg
  - 34008, Volgograd
- Serbia (5):
  - 35001, Belgrade
  - 35002, Belgrade
  - 35004, Belgrade
  - 35005, Belgrade
  - 35003, Niš
- Singapore (2):
  - 36001, Singapore
  - 36002, Singapore
- Slovenia (3):
  - 38001, Celje
  - 38003, Ljubljana
  - 38004, Novo Mesto
- South Africa (14):
  - 39003, Cape Town
  - 39016, Cape Town
  - 39017, Cape Town
  - 39011, Durban
  - 39012, Goodwood
  - 39002, Johannesburg
  - 39007, Johannesburg
  - 39010, Johannesburg
  - 39013, Johannesburg
  - 39008, Midrand
  - 39004, Port Elizabeth
  - 39006, Pretoria
  - 39014, Pretoria
  - 39019, Pretoria
- 40009, Barcelona, Spain
- Sweden (3):
  - 41001, Stockholm
  - 41004, Stockholm
  - 41002, Umeå
- Ukraine (8):
  - 43005, Crimean Autonomy
  - 43002, Dniepropetrovsk
  - 43008, Dniepropetrovsk
  - 43004, Donetsk
  - 43001, Kharkiv
  - 43007, Kiev
  - 43003, Lviv
  - 43006, Odesa

REFERENCES:
- [Background] Lichtenstein GR, Thomsen OO, Schreiber S, Lawrance IC, Hanauer SB, Bloomfield R, Sandborn WJ; Precise 3 Study Investigators. Continuous therapy with certolizumab pegol maintains remission of patients with Crohn's disease for up to 18 months. Clin Gastroenterol Hepatol. 2010 Jul;8(7):600-9. doi: 10.1016/j.cgh.2010.01.014. Epub 2010 Feb 1. PMID 20117244
- [Derived] Sandborn WJ, Wolf DC, Kosutic G, Parker G, Schreiber S, Lee SD, Abraham B, Afzali A, Arsenescu RI, Gutierrez A, Spearman M, Coarse J, Feagan BG. Effects of Transient and Persistent Anti-drug Antibodies to Certolizumab Pegol: Longitudinal Data from a 7-Year Study in Crohn's Disease. Inflamm Bowel Dis. 2017 Jul;23(7):1047-1056. doi: 10.1097/MIB.0000000000001100. PMID 28410341
- [Derived] Melmed GY, McGovern D, Schreiber S, Kosutic G, Spearman M, Coarse J, Sandborn WJ. Early remission status predicts long-term outcomes in patients with Crohn's disease treated with certolizumab pegol. Curr Med Res Opin. 2016 Dec;32(12):1937-1941. doi: 10.1080/03007995.2016.1221802. Epub 2016 Aug 22. PMID 27494777
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study started to enroll subjects in July 2004 in order to end up with 206 centers in 29 countries with enrolled subjects.
  Participant Flow refers to the Safety Population, including all enrolled subjects who received at least one injection of study treatment in feeder study C87031 [NCT00152490] or C87032 [NCT00152425].
Pre-assignment Details: All subjects who completed the Week 26 assessment in feeder studies C87031 and C87032 were eligible to enter this open-label follow-on study C87033.
Groups:
- Certolizumab Pegol: 400 mg subcutaneous injection every 4 weeks from Week 2 to Week 362.
  Certolizumab Pegol (CDP870) : Liquid for subcutaneous injection, 200 mg/ml. 400 mg at Week 2, and every 4 weeks thereafter until Week 362. Up to 84 months of therapy in this study.
Period: Overall Study
Arm/Group | Certolizumab Pegol
Started | 595 (One subject was enrolled erroneously and has no data in the database.)
Completed | 117
Not Completed | 478
Not completed — Adverse Event | 119
Not completed — Adverse Event and Other | 94
Not completed — Protocol Violation | 16
Not completed — Protocol Violation and Other | 2
Not completed — Withdrawal by Subject | 141
Not completed — Withdrawal by Subject and Other | 17
Not completed — Physician Decision | 27
Not completed — Physician Decision and Other | 6
Not completed — Lost to Follow-up | 13
Not completed — Lost to Follow-up and Other | 1
Not completed — Lack of Efficacy | 21
Not completed — Lack of Efficacy and Other | 1
Not completed — Other | 20

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Population, including all enrolled subjects who received at least one injection of study treatment in feeder study C87031 [NCT00152490] or C87032 [NCT00152425].
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 595
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 574
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 307
  Male | 288
Region of Enrollment [Number; unit: participants]
  Belarus | 12
  United States | 98
  Serbia | 29
  Estonia | 4
  Hong Kong | 2
  Spain | 1
  Ukraine | 18
  Israel | 13
  Russian Federation | 22
  Italy | 14
  Denmark | 21
  Australia | 30
  South Africa | 45
  Latvia | 4
  Slovenia | 15
  Lithuania | 1
  Austria | 4
  Czech Republic | 54
  Hungary | 48
  Canada | 17
  Belgium | 6
  Poland | 72
  Singapore | 2
  Georgia | 1
  Bulgaria | 20
  Germany | 21
  Norway | 7
  New Zealand | 10
  Sweden | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With at Least One Adverse Event (AE) During the Duration of the Study CDP870-033 (up to 84 Months)
Description: An AE is defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Time Frame: Up to 84 months from Study Entry (Week 0) to the Study End (Week 364) and the Safety Follow-up (Week 374)
Population: All 595 subjects in the Safety Population are included in the analysis of this outcome measure. Safety Population includes all enrolled subjects who received at least one injection of study treatment in feeder study C87031 [NCT00152490] or C87032 [NCT00152425].
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 595
percentage of subjects | 88.2

2. Primary Outcome: Percentage of Subjects With at Least One Serious Adverse Event (SAE) During the Duration of This Study CDP870-033 (up to 84 Months)
Description: An SAE is defined as any untoward medical occurrence that occurs at any dose which results in death, is life threatening, requires hospitalization, results in persistent/significant disability/incapacity, is an infection that requires parenteral antibiotics, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: Up to 84 months from Study Entry (Week 0) to the Study End (Week 364) and the Safety Follow-up (Week 374)
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 595
percentage of subjects | 40.3

3. Secondary Outcome: Percentage of Subjects Achieving Harvey Bradshaw Index (HBI) Remission (HBI ≤ 4) at Study Completion Visit or (Early) Withdrawal Visit
Description: HBI remission is defined as total HBI score of 4 points or less. HBI score consists of clinical parameters of general well-being (0 to 4), abdominal pain (0 to 3), number of liquid stools per day, abdominal mass (0 to 3), and complications (8 items, score 1 per item) lower scores indicating better well being. The first three parameters are scored for the previous day.
Time Frame: Study Completion Visit (Week 364) / (Early) Withdrawal Visit
Population: Of the 594 subjects in the Intention-To-Treat (ITT) Population, 592 subjects are included in the analysis of this outcome measure. ITT Population includes all subjects of the Safety Population who provide at least one efficacy measurement after Week 0 of this study.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 592
percentage of subjects | 54.7 [50.7 to 58.7]

4. Secondary Outcome: Percentage of Subjects in Harvey Bradshaw Index (HBI) Response (HBI Change >=3) at Study Completion Visit or (Early) Withdrawal Visit From Week 0 of Feeder Study CDP870-031 or CDP870-032
Description: Response is defined as decrease in total Harvey Bradshaw Index (HBI) score of 3 or more points. HBI score consists of clinical parameters of general well-being (0 to 4), abdominal pain (0 to 3), number of liquid stools per day, abdominal mass (0 to 3), and complications (8 items, score 1 per item) lower scores indicating better well-being. The first three parameters are scored for the previous day.
Time Frame: From Week 0 of study CDP870-031 [NCT00152490] or CDP870-032 [NCT00152425] to Study Completion Visit (Week 364) of this study (up to 90 months) or (Early) Withdrawal Visit
Population: All 594 subjects in the Intention-To-Treat (ITT) Population are included in the analysis of this outcome measure. ITT Population includes all subjects of the Safety Population who provide at least one efficacy measurement after Week 0 of this study.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 594
percentage of subjects | 21.7 [18.4 to 25.0]

5. Secondary Outcome: Plasma Concentration of Certolizumab Pegol at Study Completion Visit or (Early) Withdrawal Visit
Description: Plasma samples for determination of Certolizumab Pegol were taken prior to Certolizumab Pegol administration.
Time Frame: Study Completion Visit (Week 364) / (Early) Withdrawal Visit
Population: Of the 595 subjects in the Safety Population, 590 subjects are included in the analysis of this outcome measure. Safety Population includes all enrolled subjects who received at least one injection of study treatment in feeder study C87031 [NCT00152490] or C87032 [NCT00152425].
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 590
μg/mL | 5.578 [4.898 to 6.352]

6. Secondary Outcome: Percentage of Subjects With Positive Anti-CZP Anti-body Status at Any Time From Week 0 of the Feeder Study CDP870-031 or CDP870-032 to the Study Completion Visit in CDP870-033
Description: Subjects are counted as antibody positive to Certolizumab Pegol if they have at least one positive result from Week 0 in one of the previous studies CDP870-031 [NCT00152490] or CDP870-032 [NCT00152425] to the Last Visit in this study. A positive result is defined as Anti-CZP antibody levels > 2.4 units/mL.
Time Frame: From Week 0 of study CDP870-031 [NCT00152490] or CDP870-032 [NCT00152425] to Study Completion Visit (Week 364) of CDP870-033 (up to 90 months)
Population: Of the 595 subjects in the Safety Population, 593 subjects are included in the analysis of this outcome measure. Safety Population includes all enrolled subjects who received at least one injection of study treatment in feeder study C87031 [NCT00152490] or C87032 [NCT00152425].
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 593
percentage of subjects | 22.6

7. Secondary Outcome: C-Reactive Protein (CRP) Level at Study Completion Visit or (Early) Withdrawal Visit
Time Frame: Study Completion Visit (Week 364) / (Early) Withdrawal Visit
Population: Of the 594 subjects in the Intention-To-Treat (ITT) Population, 593 subjects are included in the analysis of this outcome measure. ITT Population includes all subjects of the Safety Population who provide at least one efficacy measurement after Week 0 of this study.
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 593
mg/L | 7.93 [7.14 to 8.81]

8. Secondary Outcome: Faecal Calprotectin Level at Week 258 Visit or (Early) Withdrawal Visit, if it is Earlier Than Week 258
Time Frame: Week 258 / (Early) Withdrawal Visit, if it is earlier than Week 258
Population: Of the 594 subjects in the Intention-To-Treat (ITT) Population, 567 subjects are included in the analysis of this outcome measure. ITT Population includes all subjects of the Safety Population who provide at least one efficacy measurement after Week 0 of this study.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/g stool
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 567
μg/g stool | 302.540 [267.759 to 341.839]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected up to approximately 7 years, from Study Entry (Week 0) to the Safety Follow-up (Week 374).
Description: Adverse Events refer to the Safety Population, including all enrolled subjects who received at least one injection of study treatment in feeder study C87031 [NCT00152490] or C87032 [NCT00152425].
Arm/Group | Certolizumab Pegol
Serious Adverse Events (participants affected / at risk) | 240/595
Other Adverse Events (participants affected / at risk) | 410/595
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (N=595)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (3)
Lymphadenitis (Blood and lymphatic system disorders) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (2)
Crohn's disease (Gastrointestinal disorders) | 67 (75)
Small intestinal obstruction (Gastrointestinal disorders) | 13 (16)
Intestinal obstruction (Gastrointestinal disorders) | 10 (10)
Abdominal pain (Gastrointestinal disorders) | 9 (9)
Ileal stenosis (Gastrointestinal disorders) | 7 (7)
Perirectal abscess (Gastrointestinal disorders) | 5 (5)
Anal fistula (Gastrointestinal disorders) | 4 (5)
Pancreatitis acute (Gastrointestinal disorders) | 3 (3)
Subileus (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (3)
Gastritis (Gastrointestinal disorders) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 2 (2)
Intestinal mass (Gastrointestinal disorders) | 2 (2)
Large intestine perforation (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Rectovaginal fistula (Gastrointestinal disorders) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1)
Anal inflammation (Gastrointestinal disorders) | 1 (1)
Anal stenosis (Gastrointestinal disorders) | 1 (1)
Colonic stenosis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Intestinal fistula (Gastrointestinal disorders) | 1 (1)
Intestinal stenosis (Gastrointestinal disorders) | 1 (1)
Jejunal stenosis (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1)
Oesophageal stenosis acquired (Gastrointestinal disorders) | 1 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Peritoneal adhesions (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (5)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1)
Small intestinal stricture (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Impaired healing (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1)
Biliary cirrhosis (Hepatobiliary disorders) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1)
Gallbladder non-functioning (Hepatobiliary disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1)
Perianal abscess (Infections and infestations) | 9 (10)
Abdominal abscess (Infections and infestations) | 8 (9)
Pneumonia (Infections and infestations) | 7 (7)
Gastroenteritis (Infections and infestations) | 6 (7)
Cellulitis (Infections and infestations) | 3 (3)
Disseminated tuberculosis (Infections and infestations) | 3 (3)
Pulmonary tuberculosis (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2)
Bronchopneumonia (Infections and infestations) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 2 (2)
Postoperative abscess (Infections and infestations) | 2 (4)
Pyelonephritis (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Staphylococcal infection (Infections and infestations) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 2 (2)
Abscess (Infections and infestations) | 1 (1)
Abscess intestinal (Infections and infestations) | 1 (1)
Acute tonsillitis (Infections and infestations) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Bronchitis acute (Infections and infestations) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1)
Cellulitis orbital (Infections and infestations) | 1 (1)
Chronic tonsillitis (Infections and infestations) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Epiglottitis (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Gastroenteritis clostridial (Infections and infestations) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1)
Osteomyelitis acute (Infections and infestations) | 1 (1)
Pelvic abscess (Infections and infestations) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 1 (1)
Perineal abscess (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1)
Rectal abscess (Infections and infestations) | 1 (2)
Salpingitis (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 2 (3)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Haemothorax (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (2)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1)
Polytraumatism (Injury, poisoning and procedural complications) | 1 (1)
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 1 (1)
Post procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Autoantibody positive (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone erosion (Musculoskeletal and connective tissue disorders) | 1 (1)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolisthesis acquired (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lentigo maligna stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Spinal column stenosis (Nervous system disorders) | 2 (2)
Arachnoid cyst (Nervous system disorders) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Pregnancy on oral contraceptive (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 5 (5)
Calculus ureteric (Renal and urinary disorders) | 2 (3)
Dysuria (Renal and urinary disorders) | 1 (1)
Glomerulonephritis focal (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Renal tubular acidosis (Renal and urinary disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 3 (3)
Azoospermia (Reproductive system and breast disorders) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 1 (1)
Female genital-digestive tract fistula (Reproductive system and breast disorders) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
Ovarian disorder (Reproductive system and breast disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia totalis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Pregnancy of partner (Social circumstances) | 3 (3)
Abortion induced (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Lymphangitis (Vascular disorders) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 1 (2)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (N=595)
Anaemia (Blood and lymphatic system disorders) | 34 (43)
Crohn's disease (Gastrointestinal disorders) | 130 (189)
Abdominal pain (Gastrointestinal disorders) | 89 (152)
Diarrhoea (Gastrointestinal disorders) | 64 (85)
Nausea (Gastrointestinal disorders) | 50 (83)
Dyspepsia (Gastrointestinal disorders) | 39 (46)
Vomiting (Gastrointestinal disorders) | 33 (48)
Pyrexia (General disorders) | 56 (98)
Nasopharyngitis (Infections and infestations) | 91 (201)
Urinary tract infection (Infections and infestations) | 82 (160)
Influenza (Infections and infestations) | 72 (105)
Upper respiratory tract infection (Infections and infestations) | 63 (110)
Sinusitis (Infections and infestations) | 43 (77)
Gastroenteritis (Infections and infestations) | 41 (52)
Bronchitis (Infections and infestations) | 37 (52)
Arthralgia (Musculoskeletal and connective tissue disorders) | 70 (99)
Back pain (Musculoskeletal and connective tissue disorders) | 41 (52)
Headache (Nervous system disorders) | 60 (99)
Insomnia (Psychiatric disorders) | 30 (39)
Cough (Respiratory, thoracic and mediastinal disorders) | 35 (42)
Rash (Skin and subcutaneous tissue disorders) | 40 (51)
Hypertension (Vascular disorders) | 34 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days